CLINICAL TRIAL: NCT06501053
Title: Contact Radiotherapy for Rectal Cancer (CORRECT): a Multicenter Randomized Phase II Trial
Brief Title: Contact Radiotherapy for Rectal Cancer
Acronym: CORRECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexander Valdman (Other)
Collaborators: Uppsala University Hospital (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor-Investigator, Alexander Valdman, National Principal Investigator, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CORRECT
Record Dates: First submitted 2024-07-03; First posted 2024-07-15 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Rectal Cancer
Keywords: organ sparing; brachytherapy; radiotherapy; nonoperative
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CXB + CRT (Active Comparator): Contact x-ray brachytherapy (CXB) (90Gy/3 fractions/4 weeks) and chemoradiotherapy (CRT) 45/50 Gy (1.8/2 Gy/fraction/5 weeks) with concurrent chemotherapy using capecitabine (900 mg/m2 bid, on radiation days).
  Interventions: Radiation: Radiotherapy; Radiation: Contact x-ray brachytherapy; Drug: Chemotherapy
- CXB + SCRT (Experimental): Contact x-ray brachytherapy (CXB) (90Gy/3 fractions/4 weeks) and a short-course radiotherapy (SCRT) (25 Gy in 5 daily fractions over a total time of 1 week, treating 5 days per week, 1 fraction per day, using 5 Gy per fraction, over the maximum treatment period of eight calendar days).
  Interventions: Radiation: Short-course radiotherapy; Radiation: Contact x-ray brachytherapy

INTERVENTIONS:
Radiation: Radiotherapy — 45/50 Gy (1.8/2 Gy/fraction/5 weeks)
  Arms: CXB + CRT
Radiation: Short-course radiotherapy — 25 Gy in 5 daily fractions over a total time of 1 week, treating 5 days per week, 1 fraction per day, using 5 Gy per fraction, over the maximum treatment period of eight calendar days
  Arms: CXB + SCRT
Radiation: Contact x-ray brachytherapy — 90Gy/3 fractions/4 weeks
Drug: Chemotherapy — Capecitabine (900 mg/m2 bid, on radiation days)
  Arms: CXB + CRT

SUMMARY:
The aim of the CORRECT phase 2 study is to show non-inferiority of Contact x-ray brachytherapy (CXB) + short-course radiotherapy (SCRT) compared to the experimental arm of the OPERA trial in organ preservation for early and early intermediate rectal cancer (cT1-3abN1).

DETAILED DESCRIPTION:
The primary aim of this study is to determine whether a combination of CXB + SCRT is non-inferior to CXB + chemoradiotherapy (CRT) regarding the primary endpoint 2-year organ preservation rate. Additionally, we hypothesize that a chemotherapy-free, radiation-only experimental treatment CXB+SCRT is associated with less side-effects compared to the OPERA regime.

In the OPERA trial (Gerard et al, 2023), the CXB was delivered in combination with long-course CRT. A combination of short-course radiotherapy (SCRT) and CXB has previously been used mainly in elderly and comorbid patients not suitable for long-course chemoradiotherapy. Recently, an international multi-institution report showed good outcomes of planned organ preservation using SCRT together with contact brachytherapy boost. However, no randomized data on this combination therapy are available. There are further no trials comparing CRT+CXB and SCRT+CXB.

Study participants will be randomized to either the standard treatment consisting of CXB (90Gy/3 fractions/4 weeks) and CRT 45/50 Gy (1.8/2 Gy/fraction/5 weeks) with concurrent chemotherapy using capecitabine (900 mg/m2 bid, on radiation days) OR the experimental treatment consisting of CXB (90Gy/3 fractions/4 weeks) SCRT (25 Gy in 5 daily fractions over a total time of 1 week, treating 5 days per week, 1 fraction per day, using 5 Gy per fraction, over the maximum treatment period of eight calendar days).

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the rectum classified as:
* cT1-cT3ab, < 5 cm largest diameter and < ½ circumference (MRI staging), N0-N1 (<= 3 nodes < 8mm diameter), M0
* Performance status (ECOG) 0-1
* Operable patient
* Tumor accessible to endocavitary contact X-ray brachytherapy with a distance from the lower tumor border to the anal verge ≤10 cm
* 18 years or above
* No comorbidity preventing treatment
* Patient having read the information note and having signed the informed consent
* Follow-up possible

Exclusion Criteria:

* Inoperable patient
* T3cd, T4, T≥ 5cm, Involvement of more than half of the bowel circumference
* Distance from the lower tumor border to the anal verge >10 cm
* N2-status at diagnosis or N1 with any node>= 8 mm diameter
* Patient presenting with metastasis at diagnosis (M1)
* Previous pelvic irradiation
* Tumor with extramural vascular invasion
* Poorly differentiated tumor
* Simultaneous progressive cancer
* Tumor invading external anal sphincter or growth within 1 mm of the levator
* Tumor within 1 mm from MRF (mesorectal fascia)
* Patient unable to receive CXB or CRT
* Any significant concurrent medical illness that in the opinion of the investigator would preclude protocol therapy
* Patient with history of poor compliance or current or past psychiatric conditions or severe acute or chronic medical conditions that would interfere with the ability to comply with the study protocol
* Concurrent enrolment in another clinical trial using an investigational anti-cancer treatment within 28 days prior to the first dose of study treatment
* Total DPD deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
Rectum preservation | At 24 months after start of treatment
  Proportion of patients with successful rectum preservation after standard vs experimental treatment. Organ preservation is considered to have failed if the rectum is removed OR if the patient develops non-salvageable locoregional failure

SECONDARY OUTCOMES:
Acute treatment-related toxicity | From start of treatment until 90 days after ending treatment
  Incidence of grade 3-5 toxicity as assessed by CTCAE v5.0
Late treatment related toxicity | From 90 days after ending treatment until end of study
  Incidence of grade 3-5 toxicity as assessed by CTCAE v5.0
Clinical complete response (cCR) | At 14-16 and 24-26 weeks after start of treatment
  Proportion of patients with cCR as assessed by DRE, endoscopy, MRI-T2W, and MRI-DWI
Postoperative complications | Within the first 30 days after Total Mesorectal Excision (TME) surgery
  Difference in postoperative complications (graded according to Clavien-Dindo) after standard vs experimental treatment
Stoma | At 12 and 24 months after start of treatment
  Proportion of patients with a stoma
Metastasis-free survival | At 24 months after start of treatment
  Survival without sign of metastasis after standard vs experimental treatment
Locoregional failure | At 24 months after start of treatment
  Proportion of patients with locoregional failure after standard vs experimental treatment
Overall survival | At 24 months after start of treatment
  Overall survival after standard vs experimental treatment
TME-free survival | At 24 months after start of treatment
  Survival without Total Mesorectal Excision after standard vs experimental treatment
Salvage TME resections | From 24 weeks after start of treatment until end of study
  Rate of R0 Total Mesorectal Excisions after standard vs experimental treatment
Tumor regression grade | After 14-16 weeks and 24-26 weeks after start of treatment
  Tumor regression grade in the surgical specimen (R0, ypT0, ypTNM) after standard vs experimental treatment
Sphincter preservation | At 24 months after start of treatment
  Rate of sphincter preservation after standard vs experimental treatment
General Health Related Quality of Life (HR QoL) | At baseline and at 3, 6, 12, 24, 36, 48 and 60 months after start of treatment
  General Health Related Quality of Life (HR QoL) as measured by the European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire QLQ-C30. Responses made on a Likert scale are transformed to a score from 0 to 100 where a higher score indicate a better quality of life
Colorectal cancer specific Health Related Quality of Life (HR QoL) | At baseline and at 3, 6, 12, 24, 36, 48 and 60 months after start of treatment
  Health Related Quality of Life (HR QoL) as measured by the European Organisation for Research and Treatment of Cancer (EORTC) colorectal cancer specific quality of life questionnaire QLQ-CR29. Responses made on a Likert scale are transformed to a score from 0 to 100 where a higher score indicate a better quality of life
Bowel function | At baseline, 3, 6, 12, 24, 36, 48 and 60 months after start of treatment
  Bowel function as assessed by the Low Anterior Resection Syndrome (LARS) score. LARS is scored from 0 to 42 points and a higher score indicates worse outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Karolinska University Hospital, Theme Cancer, Dept of Pelvic cancer, Stockholm, Solna
  - Uppsala University Hospital, Colorectal Surgery, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data that underlie the reported results.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal and whose proposed use of the data has been approved by an independent review committee. A data-sharing agreement will also be required. Contact: alexander.valdman@ki.se

REFERENCES:
- [Background] Gerard JP, Barbet N, Schiappa R, Magne N, Martel I, Mineur L, Deberne M, Zilli T, Dhadda A, Myint AS; ICONE group. Neoadjuvant chemoradiotherapy with radiation dose escalation with contact x-ray brachytherapy boost or external beam radiotherapy boost for organ preservation in early cT2-cT3 rectal adenocarcinoma (OPERA): a phase 3, randomised controlled trial. Lancet Gastroenterol Hepatol. 2023 Apr;8(4):356-367. doi: 10.1016/S2468-1253(22)00392-2. Epub 2023 Feb 16. PMID 36801007
- [Derived] Nilsson PJ, Folkesson J, Marsk R, Radu C, Stratulat I, Blomqvist L, Martling A, Valdman A. Contact radiotherapy for rectal cancer (CORRECT): study protocol for a multicentre randomised phase II trial. BMJ Open. 2025 Apr 9;15(4):e100356. doi: 10.1136/bmjopen-2025-100356. PMID 40204311